CLINICAL TRIAL: NCT03041428
Title: Effect of Ultraprotective Ventilation on the Lung Inflammatory Response in Patients With Acute Pulmonary Edema Treated With Venoarterial Extracorporeal Oxygenation
Brief Title: Ultra Protective Ventilation During Venoarterial Extracorporeal Membrane Oxygenation (UPV-ECMO)
Acronym: UPV-ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FINBA_CritLab_1
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cardiogenic Pulmonary Edema; Ventilator-Induced Lung Injury; Extracorporeal Circulation; Complications
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recruited patients (Experimental): Ultraprotective ventilation
  Interventions: Device: Ultraprotective ventilation

INTERVENTIONS:
Device: Ultraprotective ventilation — Adjusting ventilator parameters for 3 ml/kg of tidal volume in order to achieve the ultra protective strategy

SUMMARY:
Mechanical ventilation, in spite of being a life-saving technique, can also induce lung injury (VILI) mediated by an inflammatory response, thus having a profound impact in the course of critically ill patients. Ventilatory strategies aimed to minimize this VILI have reduced mortality rates. Patients suffering cardiogenic pulmonary edema may need venoarterial extracorporeal oxygenation, at the same time they are being mechanically ventilated. The objective of this study is to analyze changes induced by the use of utraprotective ventilatory strategies in the inflammatory lung response of these patients and their impact on outcomes.

DETAILED DESCRIPTION:
Mechanical ventilation is the cornerstone of the critically-ill patients support, providing better gas exchange conditions while respiratory muscles rest. Providing this life-support technique may be harmful on the lung tissue, last decades research efforts were focused on minimizing the ventilator-induced lung injury (VILI). Knowledge regarding the mechanisms of this injury has led to changes in the clinical practice, consisting on the application of positive end-expiratory pressure (PEEP) and the use of low tidal volumes, giving rise to the strategy known as "protective ventilation". Moreover, the use of extracorporeal membrane oxygenation (ECMO) techniques contributes to maintaining an adequate gas exchange until lung damage resolution. A tidal volume in the range of 6 ml/Kg of ideal body weight, with a reasonable level of PEEP is the standard of care for patients with the ARDS. However, optimal levels of tidal volume and PEEP have not been completely established. On the other side, decreasing tidal volume below 6 ml/Kg faces its own problems. The role of the so-called "ultraprotective" approaches, in which extracorporeal support is required to reduce tidal volumes up to 3 ml/kg or less, although feasible, is currently under research. During venoarterial ECMO, blood is removed from the vessels and pumped through a circuit where is oxygenated and CO2 is removed; finally, the blood is returned to the arterial circulation. The development of new circuits and devices made this therapy become safer and more useful, improving outcomes so that its application has been widespread to many centers all over the world. One of the ECMO advantages is carbon dioxide removal, which allows reducing tidal volume below 6 ml/kg. Ultraprotective strategies with 3 ml/kg have demonstrated to be feasible, but the additional benefit of this strategy is to be demonstrated. Therefore, in this study, patients suffering cardiogenic pulmonary edema requiring ECMO and mechanical ventilation are submitted to an ultraprotective ventilator strategy. Lung inflammatory response is measured before and after the intervention, in order to evaluate its impact in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic pulmonary edema supported by venoarterial extracorporeal membrane oxygenation.
* Invasive mechanical ventilatory support under sedation.

Exclusion Criteria:

* Immunosupresion.
* Hemodynamic instability refractory to mechanical support, conditioning an end-of-life approach and terminal situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in lung inflammatory mediators levels | Baseline and 18 hours after the intervention
  Bronchoalveolar lavage cytokines levels, measured in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Albaiceta, Principal Investigator — HUCA-FINBA, Universidad de Oviedo
Locations (1):
- Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Yes
All datasets underlying the study are available upon request to the study principal investigators. All of the individual participant data collected during the trial, informed consent forms, study protocol, statistical analysis plan, analytic R code and raw data, are available under reasonable request, and after deindentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 3 months after publication.
Access Criteria: Principal investigators will review requests of data to be provided.

REFERENCES:
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Leligdowicz A, Fan E. Extracorporeal life support for severe acute respiratory distress syndrome. Curr Opin Crit Care. 2015 Feb;21(1):13-9. doi: 10.1097/MCC.0000000000000170. PMID 25517890
- [Background] Determann RM, Royakkers A, Wolthuis EK, Vlaar AP, Choi G, Paulus F, Hofstra JJ, de Graaff MJ, Korevaar JC, Schultz MJ. Ventilation with lower tidal volumes as compared with conventional tidal volumes for patients without acute lung injury: a preventive randomized controlled trial. Crit Care. 2010;14(1):R1. doi: 10.1186/cc8230. Epub 2010 Jan 7. PMID 20055989
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Background] Figueroa-Casas JB, Montoya R. Effect of Tidal Volume Size and Its Delivery Mode on Patient-Ventilator Dyssynchrony. Ann Am Thorac Soc. 2016 Dec;13(12):2207-2214. doi: 10.1513/AnnalsATS.201605-362OC. PMID 27598383
- [Background] Bein T, Weber-Carstens S, Goldmann A, Muller T, Staudinger T, Brederlau J, Muellenbach R, Dembinski R, Graf BM, Wewalka M, Philipp A, Wernecke KD, Lubnow M, Slutsky AS. Lower tidal volume strategy ( approximately 3 ml/kg) combined with extracorporeal CO2 removal versus 'conventional' protective ventilation (6 ml/kg) in severe ARDS: the prospective randomized Xtravent-study. Intensive Care Med. 2013 May;39(5):847-56. doi: 10.1007/s00134-012-2787-6. Epub 2013 Jan 10. PMID 23306584
- [Background] Fan E, Gattinoni L, Combes A, Schmidt M, Peek G, Brodie D, Muller T, Morelli A, Ranieri VM, Pesenti A, Brochard L, Hodgson C, Van Kiersbilck C, Roch A, Quintel M, Papazian L. Venovenous extracorporeal membrane oxygenation for acute respiratory failure : A clinical review from an international group of experts. Intensive Care Med. 2016 May;42(5):712-724. doi: 10.1007/s00134-016-4314-7. Epub 2016 Mar 23. PMID 27007108
- [Background] Schmidt M, Stewart C, Bailey M, Nieszkowska A, Kelly J, Murphy L, Pilcher D, Cooper DJ, Scheinkestel C, Pellegrino V, Forrest P, Combes A, Hodgson C. Mechanical ventilation management during extracorporeal membrane oxygenation for acute respiratory distress syndrome: a retrospective international multicenter study. Crit Care Med. 2015 Mar;43(3):654-64. doi: 10.1097/CCM.0000000000000753. PMID 25565460
- [Derived] Amado-Rodriguez L, Del Busto C, Lopez-Alonso I, Parra D, Mayordomo-Colunga J, Arias-Guillen M, Albillos-Almaraz R, Martin-Vicente P, Lopez-Martinez C, Huidobro C, Camporota L, Slutsky AS, Albaiceta GM. Biotrauma during ultra-low tidal volume ventilation and venoarterial extracorporeal membrane oxygenation in cardiogenic shock: a randomized crossover clinical trial. Ann Intensive Care. 2021 Aug 28;11(1):132. doi: 10.1186/s13613-021-00919-0. PMID 34453620